CLINICAL TRIAL: NCT03856489
Title: Patients' Sleep at the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-10-SLEEP
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Sleep Quality of ICU Patients
Keywords: sleep; intensive care unit; patient; nurse; inter-rater reliability; Richards-Campbell sleeping questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: This study group will consist of patients hospitalized at ICU, who will be given the Richards-Campbell Sleeping Questionnaire (RCSQ) to fill in every morning between 7 am and 10 am.
  Interventions: Other: Richards-Campbell Sleeping Questionnaire (RCSQ)
- Nurses: This study group will consist of patients hospitalized at ICU, who will be given the Richards-Campbell Sleeping Questionnaire (RCSQ) to fill in every morning between 7 am and 7:30 am.
  Interventions: Other: Richards-Campbell Sleeping Questionnaire (RCSQ)

INTERVENTIONS:
Other: Richards-Campbell Sleeping Questionnaire (RCSQ) — This five-item visual analogue scale was designed as an outcome measure for assessing the perception of sleep in critically ill patients. The scale evaluates perceptions of depth of sleep, sleep onset latency, number of awakenings, time spent awake, and overall sleep quality.

SUMMARY:
The primary objective of this study is to evaluate patient-nurse reliability and agreement of the Richards-Campbell sleep questionnaire (RCSQ) in a population of medical intensive care unit patients.

DETAILED DESCRIPTION:
The main instrument of this research is the Richards Campbell Sleeping Questionnaire (RCSQ) regarding patients' overnight sleep quality. This questionnaire is given to complete to eligible patients between 7 am and 10 am. The same questionnaire is given to the night-shift nurse between 7 am and 7:30 am, who was taking care of that particular patient overnight. This RCQS assessment is based solely on each nurse´s perception of the patient´s sleep quality last night. Neither the nurse nor the patient know each other´s RCSQ response.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients
* Age 18 years and older
* Glasgow coma scale 15

Exclusion Criteria:

* Age < 18 years
* Glasgow coma scale < 15

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at intensive care units at the University Hospital Ostrava, Czech Republic fulfiling the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Patient-nurse inter-rater reliability | 30 weeks
  The inter-rater reliability between the evaluation of sleep quality performed by the patient and the nurse, as per Richards-Campbell Sleeping Questionnaire (RCSQ) score achieved, will be assessed. The RCSQ tool is used to assess a total of five dimensions pertaining to sleep, each of which is evaluated on a scale of 0 to 100.

SECONDARY OUTCOMES:
Patient sleep quality | 30 weeks
  The quality of patient sleep will be evaluated using the achieved Richards-Campbell Sleeping Questionnaire (RCSQ) scores. The RCSQ tool is used to assess a total of five dimensions pertaining to sleep, each of which is evaluated on a scale of 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Tejkalová, Mgr., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to make individual participant data available to other researchers.

REFERENCES:
- [Background] Kamdar BB, Shah PA, King LM, Kho ME, Zhou X, Colantuoni E, Collop NA, Needham DM. Patient-nurse interrater reliability and agreement of the Richards-Campbell sleep questionnaire. Am J Crit Care. 2012 Jul;21(4):261-9. doi: 10.4037/ajcc2012111. PMID 22751369
- [Background] Frisk U, Nordstrom G. Patients' sleep in an intensive care unit--patients' and nurses' perception. Intensive Crit Care Nurs. 2003 Dec;19(6):342-9. doi: 10.1016/s0964-3397(03)00076-4. PMID 14637294